CLINICAL TRIAL: NCT00673777
Title: Phase I/II Study of Multiple-Vaccine Therapy Using Epitope Peptide Restricted to HLA-A*0201 in Treating Patients With Refractory Non-Small Cell Lung Cancer
Brief Title: Histocompatibility Leukocyte Antigen (HLA)-A*0201 Restricted Peptide Vaccine Therapy in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Infectious Disease and Applied Immunology, The Institute of Medical Science, The University of Tokyo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMS-NSCLC02
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: HLA-A*0201; Peptide Vaccine; URLC10; VEGFR1; VEGFR2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — LY6K protein, human; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: URLC10, VEGFR1 and VEGFR2

INTERVENTIONS:
Biological: URLC10, VEGFR1 and VEGFR2 — Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, the URLC10-117 peptide(1mg), VEGFR1 peptide(1mg) and VEGFR2 peptide(1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection.

SUMMARY:
The purpose of this study is to evaluate the safety and time to progression of HLA-A*0201 restricted epitope peptides URLC10, VEGFR1 and VEGFR2 emulsified with Montanide ISA 51.

DETAILED DESCRIPTION:
URLC10 has been identified as cancer specific molecules especially in non small cell lung cancer using genome-wide expression profile analysis by cDNA microarray technique. We have determined the HLA-A*0201 restricted epitope peptides derived from these molecules. We also tend to use the peptides targeting to tumor angiogenesis. VEGF receptor 1 and 2 are essential targets to tumor angiogenesis, and we identified that peptides derived from these receptors significantly induce the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of those peptides. Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, the URLC10-117 peptide(1mg), VEGFR1 peptide(1mg) and VEGFR2 peptide(1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection. Repeated cycles of vaccine will be administered until patients develop progressive disease or unacceptable toxicity, whichever occurs first. In the phase I study, we evaluate the safety and tolerability of these peptide vaccine. In the following phase II study, we evaluate the immunological and clinical response of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

Disease characteristics

* Advanced or recurrent non small cell lung cancer
* Second line or later therapeutic status Patient characteristics
* ECOG performance status 0-2
* Life expectancy > 3 months
* HLA-A*0201
* Laboratory values as follows

  * 2000/mm3<WBC<15000/mm3
  * Platelet count>100000/mm3
  * Bilirubin < 3.0mg/dl
  * Asparate transaminase < 150IU/L
  * Alanine transaminase < 150IU/L
  * Creatinine < 3.0mg/dl
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception)
* Breastfeeding
* Active or uncontrolled infection
* Unhealed external wound
* Concurrent treatment with steroids or immunosuppressing agent
* Prior chemotherapy,radiation therapy, or immunotherapy within 4 weeks
* Uncontrolled brain and/or intraspinal metastasis
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
safety(Phase I:toxicities as assessed by NCI CTCAE version3) and efficacy(Phase II:Feasibility as evaluated by RECIST) | two months

SECONDARY OUTCOMES:
To evaluate immunological responses | two months
Time to progression | one years

CONTACTS AND LOCATIONS:
Overall Officials: Naohida Yamashita, MD/PhD, Study Chair — Tokyo University
Locations (1):
- The Institute of Medical Science, The University of Tokyo, Tokyo, Tokyo, Japan

REFERENCES:
- [Background] Suda T, Tsunoda T, Uchida N, Watanabe T, Hasegawa S, Satoh S, Ohgi S, Furukawa Y, Nakamura Y, Tahara H. Identification of secernin 1 as a novel immunotherapy target for gastric cancer using the expression profiles of cDNA microarray. Cancer Sci. 2006 May;97(5):411-9. doi: 10.1111/j.1349-7006.2006.00194.x. PMID 16630140
- [Background] Daigo Y, Nakamura Y. From cancer genomics to thoracic oncology: discovery of new biomarkers and therapeutic targets for lung and esophageal carcinoma. Gen Thorac Cardiovasc Surg. 2008 Feb;56(2):43-53. doi: 10.1007/s11748-007-0211-x. Epub 2008 Feb 24. PMID 18297458
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261